CLINICAL TRIAL: NCT03505242
Title: Bronchial Blocker in Blocking the Right Middle Lower Lobe Versus Double-Lumen Endotracheal Tube for One-Lung Ventilation in Minimally Invasive Cardiac Surgery
Brief Title: Application of Bronchial Blocker in Minimally Invasive Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABMICS
Record Dates: First submitted 2017-08-30; First posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Minimally Invasive Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BB (Experimental)
  Interventions: Device: bronchial blocker for BB group
- DLT (Experimental)
  Interventions: Device: double lumen tube for DLT group

INTERVENTIONS:
Device: bronchial blocker for BB group — Using bronchial blocker to block right middle lower lobe during surgery.
  Arms: BB
Device: double lumen tube for DLT group — Using double lumen tube to achieve single lung ventilation during surgery.
  Arms: DLT

SUMMARY:
Both left single lung ventilation by left double lumen tube and bilateral ventilation with selective blockage of right middle lower lobe by bronchial blocker can provide suitable surgical field for minimally invasive cardiac surgery. The current study was designed to compare the impact of these two different methods on oxygenation, degree of pulmonary collapse and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-III
* BMI 18-31
* elective minimally invasive cardiac surgery by right thoracotomy

Exclusion Criteria:

* asthma
* COPD
* previous lung surgery
* previous cardiac surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
oxygenation | intraoperative
  record SpO2 and PaO2 during selective ventilation

SECONDARY OUTCOMES:
degree of pulmonary collapse | intraoperative
  surgeon score the degree of pulmonary collapse (1 for no pulmonary collapse and 5 for excellent pulmonary collapse)

IPD SHARING:
Plan to Share IPD: No